CLINICAL TRIAL: NCT01279421
Title: High Risk Crack Use Settings and HIV in El Salvador
Acronym: Encuentro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Julia Dickson-Gomez, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00013931; R01DA020350 (NIH)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: HIV; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social Network HIV Testing (Experimental): Participants in this arm will be recruited through social networks and will receive an HIV test.
  Interventions: Behavioral: Social Network HIV Testing
- Peer Network Intervention (Experimental): Eight (8) current or former crack users will be recruited to facilitate small networks of crack users in a three-day intervention. They will also facilitate monthly meetings open to all community members regarding HIV prevention and interpersonal violence.
  Interventions: Behavioral: Peer Network Intervention

INTERVENTIONS:
Behavioral: Social Network HIV Testing — Crack users will be recruited for HIV testing and receive 3 coupons to recruit other crack users for HIV testing.
  Arms: Social Network HIV Testing
Behavioral: Peer Network Intervention — Peer leaders will recruit small networks of crack users and facilitate a three-day prevention intervention.
  Arms: Peer Network Intervention

SUMMARY:
This project will first increase the accessibility and acceptability of rapid HIV testing in health clinics located in or near four low-income communities in San Salvador, El Salvador. The investigators will use crack users' social networks and small incentives, as recommended by the CDC, in collaboration with the Salvadoran Ministry of Public Health and Social Assistance (MSPAS) to encourage crack users to receive HIV testing. The second part of the intervention consists of training 8 Peer Leaders to recruit and lead a Peer Network Intervention among 400 crack users to change norms supporting HIV protective behaviors. The intervention will include monthly meetings open to crack using and non-crack using community residents to reinforce HIV risk reduction skills, and discussion of other topics related to HIV such as illicit drug use and interpersonal violence and community-wide HIV awareness events. Our hypothesis is that these two intervention features will singly, and in combination, reduce HIV risk behaviors among Salvadoran crack users.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* used crack cocaine in the last 2 weeks

Exclusion Criteria:

* not giving informed consent
* under 18 years of age
* considered by research staff to be unfit or unable to give informed consent
* engages in continued disruptive behavior while participating in the project
* not using crack or cocaine in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4382 (Actual)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Increased HIV testing rates among crack users | 24 months
Decreased number of sexual risk behaviors among crack users | 12 months

SECONDARY OUTCOMES:
Community and organizational factors associated with successful implementation of multi-level, community-based HIV prevention intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia B. Dickson-Gomez, Ph.D., Principal Investigator — Medical College of Wisconsin; Gloria Bodnar, Ph.D., Study Director — Fundacion Antidrogas de El Salvador (FUNDASALVA)
Locations (1):
- Fundasalva, San Salvador, El Salvador

REFERENCES:
- [Background] Dickson-Gomez J, Bodnar G, Petroll A, Johnson K, Glasman L. HIV Treatment for Alcohol and Non-Injection Drug Users in El Salvador. Qual Health Res. 2015 Dec;25(12):1719-32. doi: 10.1177/1049732314568322. Epub 2015 Jan 16. PMID 25595149
- [Background] Dickson-Gomez J, Corbett AM, Bodnar G, Zuniga MO, Guevara CE, Rodriguez K, Navas V. Context and group dynamics in a CBPR-developed HIV prevention intervention. Health Promot Int. 2016 Mar;31(1):93-105. doi: 10.1093/heapro/dau058. Epub 2014 Jul 28. PMID 25070835
- [Background] Dickson-Gomez J. Substance abuse disorders treatment in El Salvador: analysis of policy-making-related failure. Subst Use Misuse. 2012 Nov-Dec;47(13-14):1546-51. doi: 10.3109/10826084.2012.705698. PMID 23186469
- [Background] Dickson-Gomez J, McAuliffe T, Rivas de Mendoza L, Glasman L, Gaborit M. The relationship between community structural characteristics, the context of crack use, and HIV risk behaviors in San Salvador, El Salvador. Subst Use Misuse. 2012 Feb;47(3):265-77. doi: 10.3109/10826084.2011.635325. PMID 22217125
- [Background] Dickson-Gomez J, Bodnar G, Guevara CE, Rodriguez K, De Mendoza LR, Corbett AM. With God's help i can do it: crack users? Formal and informal recovery experiences in El Salvador. Subst Use Misuse. 2011;46(4):426-39. doi: 10.3109/10826084.2010.495762. Epub 2010 Aug 24. PMID 20735191
- [Background] Dickson-Gomez J. Structural factors influencing patterns of drug selling and use and HIV risk in the San Salvador metropolitan area. Med Anthropol Q. 2010 Jun;24(2):157-81. doi: 10.1111/j.1548-1387.2010.01095.x. PMID 20550091
- [Background] Dickson-Gomez J, Corbett AM, Bodnar G, Rodriguez K, Guevara CE. Resources and obstacles to developing and implementing a structural intervention to prevent HIV in San Salvador, El Salvador. Soc Sci Med. 2010 Feb;70(3):351-359. doi: 10.1016/j.socscimed.2009.10.029. Epub 2009 Nov 10. PMID 19910099
- [Result] Glasman LR, Dickson-Gomez J, Lechuga J, Tarima S, Bodnar G, de Mendoza LR. Using Peer-Referral Chains with Incentives to Promote HIV Testing and Identify Undiagnosed HIV Infections Among Crack Users in San Salvador. AIDS Behav. 2016 Jun;20(6):1236-43. doi: 10.1007/s10461-015-1267-8. PMID 26687093